CLINICAL TRIAL: NCT00389779
Title: A Phase 3 Randomized, Double-Blind, Placebo- and Active-Controlled, Multi-center, Parallel Group Study to Evaluate the Safety and Efficacy of Darusentan in Subjects With Resistant Hypertension Receiving Combination Therapy With Three or More Antihypertensive Drugs, Including a Diuretic, as Compared to Guanfacine or Placebo (Protocol DAR-312)
Brief Title: DORADO-AC - Optimized Doses of Darusentan as Compared to an Active Control in Resistant Hypertension
Acronym: Darusentan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol DAR-312
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — darusentan; Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Darusentan (Experimental): Placebo to match darusentan for 2-week placebo run-in period, followed by darusentan capsules titrated to an optimal dose of 50 mg, 100 mg, or 300 mg administered orally once daily for 14 weeks
  Interventions: Drug: Darusentan; Drug: Darusentan Placebo
- Guanfacine (Active Comparator): Placebo to match darusentan for 2-week placebo run-in period, followed by guanfacine 1 mg capsules administered orally once daily for 14 weeks
  Interventions: Drug: Guanfacine; Drug: Darusentan Placebo
- Darusentan Placebo (Placebo Comparator): Placebo to match darusentan for 2-week placebo run-in period, followed by placebo to match darusentan administered orally once daily for 14 weeks
  Interventions: Drug: Darusentan Placebo

INTERVENTIONS:
Drug: Darusentan — Darusentan capsules administered orally once daily
  Other Names: LU 135252
  Arms: Darusentan
Drug: Guanfacine — Guanfacine capsules administered orally once daily
  Arms: Guanfacine
Drug: Darusentan Placebo — Placebo to match darusentan administered orally once daily

SUMMARY:
This is a randomized, double-blind, placebo- and active-controlled study of a new experimental drug called darusentan. Darusentan is not currently approved by the United States Food and Drug Administration (FDA), which means that a doctor cannot prescribe this drug. The purpose of this study is to determine if darusentan is effective in reducing systolic and diastolic hypertension despite treatment with full doses of three or more antihypertensive drugs, including a diuretic. Subjects will be randomized to darusentan (optimized dose), an active comparator, or placebo, administered orally. The treatment period for this trial is 14 weeks.

ELIGIBILITY:
SELECTED INCLUSION CRITERIA:

1. Subjects who are competent to provide written consent;
2. Aged 35 to 80 years;
3. Subjects with diabetes and/or chronic kidney disease must have an average sitting systolic blood pressure greater than or equal to 130 mmHg;
4. All other subjects must have an average sitting systolic blood pressure greater than or equal to 140 mmHg;
5. Receiving and adhering to full doses of appropriate guideline-recommended antihypertensive drugs from three different classes of antihypertensive agents, including a diuretic;
6. Female subjects of non-childbearing potential (i.e., post-menopausal for at least 2 years or surgically sterile).

SELECTED EXCLUSION CRITERIA:

1. Average sitting systolic and diastolic blood pressure greater than or equal to 180 mmHg and 110 mmHg, respectively;
2. Subjects treated with a central alpha-2 agonist and/or imidazoline receptor agonist;
3. Left ventricular dysfunction;
4. Serum ALT or AST greater than 2 times the Upper Limit of Normal;
5. Subjects who have experienced myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months; or sick sinus syndrome or second or third degree atrioventricular block, atrial fibrillation or recurrent atrial tachycardia, recurrent ventricular tachycardia, or symptomatic bradycardia;
6. Implanted pacemakers or cardioverter defibrillator;
7. Symptomatic congestive heart failure requiring treatment;
8. Hemodynamically significant valvular heart disease;
9. Hemodialysis or peritoneal dialysis, or history of renal transplant;
10. Type I diabetes mellitus;
11. Diagnosis or recurrence of malignancy within the past 3 years;
12. Sleep apnea, unless a recent sleep study demonstrated arterial oxygenation saturation greater than or equal to 90%, treated or untreated;
13. Subjects who perform alternating shift or night work;
14. Subjects who have participated in a clinical study involving another investigational drug or device within 4 weeks prior to Screening

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough sitting systolic and diastolic blood pressure measured by sphygmomanometry | Baseline to Week 14

SECONDARY OUTCOMES:
Percentage of subjects reaching systolic blood pressure goal after 14 weeks of treatment | Week 14
Change from baseline in mean 24-hour systolic and diastolic blood pressure measured by ambulatory blood pressure monitoring (ABPM) | Baseline to Week 14
Change from baseline in estimated glomerular filtration rate (eGFR) | Baseline to Week 14

CONTACTS AND LOCATIONS:
Locations (146):
- United States (86):
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - The Heart Center, PC, Huntsville, Alabama
  - Mulberry Medical Associates, PC, Montgomery, Alabama
  - Arizona Center for Clinical Research, Glendale, Arizona
  - Cardiovascular Consultants, Ltd., Glendale, Arizona
  - Lovelace Scientific Resources, Inc, Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Southwest Heart, Tucson, Arizona
  - HealthFirst Physician of AR, PA dba Convenient Care Clinic, Hot Springs, Arkansas
  - NEA Clinic, Jonesboro, Arkansas
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Medical Investigations Inc., Little Rock, Arkansas
  - Highgrove Medical Center, Bakersfield, California
  - Central Cardiology Medical Clinic, Bakersfield, California
  - Impact Clinical Trials, Beverly Hills, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Pacific Heart Institute, Santa Monica, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Doctors Medical Center of Walton County, DeFuniak Springs, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Maxine Hamilton, MD, PA, Fort Lauderdale, Florida
  - St. John's Center for Clinical Research, Jacksonville, Florida
  - Private Practice of Dr. Bridget Bellingar, Largo, Florida
  - A+ Research Inc., Miami, Florida
  - AppleMed Research, Inc., Miami, Florida
  - Internal Medicine Associates of South Florida, North Miami Beach, Florida
  - Ormond Medical Arts Pharmaceutical Research center, Ormond Beach, Florida
  - Northwest Florida Heart Group, PA - Research Dept, Pensacola, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Suncoast Cardiovascular Research, Inc., St. Petersburg, Florida
  - Tampa Bay Nephrology Associates, PL, Tampa, Florida
  - Orlando Rangel, MD, PA, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - AMR Research Associates, LLC, Bogart, Georgia
  - Atlanta Vascular Research Foundation, Tucker, Georgia
  - North Shore Cardiologist, Bannockburn, Illinois
  - Consultants in Cardiovascular Med (CIS), Melrose Park, Illinois
  - Illinois Heart & Lunch Research, Normal, Illinois
  - Methodist Medical Center-Heart, Lung & Vascular Institute, Peoria, Illinois
  - Medical Consultants, PC, Muncie, Indiana
  - University Medical Associates, Louisville, Kentucky
  - Dr. Jeffrey Chen, Lafayette, Louisiana
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - Maine Research Associate, Auburn, Maine
  - PrimeCare Internal Medicine, Biddeford, Maine
  - Great Lakes Heart Center of Alpena, Alpena, Michigan
  - Internal Medicine of Nothern Michigan, Petoskey, Michigan
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Central Minnesota Heart Center at St. Cloud Hospital, Saint Cloud, Minnesota
  - St. Paul Cardiology, Saint Paul, Minnesota
  - Glacier View Cardiology, PC, Kalispell, Montana
  - Impact Clinical Trials, Las Vegas, Nevada
  - NJ Heart, Linden, New Jersey
  - New Jersey Physicians, Passaic, New Jersey
  - Lifeline Research Institute, Brooklyn, New York
  - Metrolina Internal Medicine, PA, Charlotte, North Carolina
  - Heart Care Center of Charlotte, Charlotte, North Carolina
  - Physicians East, PA, Winterville, North Carolina
  - Plaza Medical Group, PC, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Counsultants, LLC, Tulsa, Oklahoma
  - Integrated Medical Research PC, Ashland, Oregon
  - Blackstone Cardiology Associates, Pawtucket, Rhode Island
  - Charleston Cardiology, Charleston, South Carolina
  - Paris View Family Practice, Greenville, South Carolina
  - Internal Medicine of Greer, Greer, South Carolina
  - Scenic City Research, Cleveland, Tennessee
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Cardiovascular Research Inst. of Dallas, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Sergio F Rovner, MD, El Paso, Texas
  - Salim Gopalani, MD, PA, Houston, Texas
  - Humayun Mirza, MD, PA, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Houston Clinical Research Assoc., Houston, Texas
  - Innovative Research of West Florida, Hurst, Texas
  - North Texas Medical Research, Plano, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Fletcher Allen Health Care/University of Vermont, Burlington, Vermont
  - Kamlesh N. Dave Cardiology, Hopewell, Virginia
  - WVU Physicians of Charleston, Charleston, West Virginia
  - Alpha Medical Research, LLC, Madison, Wisconsin
  - Executive Health and Research Associates, Madison, Wisconsin
- Argentina (15):
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Consultorios Medicos Privados S.A., Buenos Aires
  - Hospital General de Agudos "Dr. Abel Zubizarreta", Buenos Aires
  - Policlinica Bancaria "9 de Julio", Buenos Aires
  - Diabaid (Instituto de Asistencia Integral en Diabetes), Ciudad de Buenos Aires
  - MD Investigaciones, Ciudad de Buenos Aires
  - Centro Medico Privado, Ciudad de
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Fundacion Rusculleda, Córdoba
  - Framingham Centro Medico, La Plata
  - Instituto de Investigaciones Clinicas de Quilmes, Quilmes
  - Instituto de Investigaciones Clinicas, Rosario
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Australia (4):
  - Flinders Medical Centre, Bedford Park
  - Royal Brisbane & Women's Hospital, Herston
  - Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
- Belgium (11):
  - U.Z. Brussel, Brussels
  - Private Practice of Dr. Geert Hollanders, De Pinte
  - Private Practice of Dr. Francis Vrancken, Genk
  - Private Practice of Dr. Herwig Van Aerde, Genk
  - Private Practice of Dr. Willy Denier, Genk
  - Private Practice of Dr. Herman Docx, Hoeilaart
  - Private Practice of Dr. Yohan Balthazar, Natoye
  - Private Practice of Dr. Sophie Baeyens, Pulle
  - Private Practice of Dr. Jean Gilissen, Riemst
  - Private Practice of Dr. Guido Mehuys, Tielt
  - Private Practice of Dr. Luc Capiau, Wetteren
- Hospital Universitario Pedro Ernesto, Rio de Janeiro, Brazil
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Region Sjaelland, Storstrommens Sygenhus, Naestved, Næstved
- France (10):
  - Private Practice of dr. Marty Jacques, Mûrs-Erigné, Murs-Erigne
  - George Delamare, Blois
  - Centre d'Investigation Clinique, Dommartin-lès-Toul
  - Private Practice of Dr. Brune Charrier, La Jubaudière
  - Private Practice of Dr. Jean Boulet-Gercourt, Le Mesnil-en-Vallée
  - Private Practice of Dr. Gildas Ganuchaud, Le Temple-de-Bretagne
  - Private Practice of Dr. Jacques Samat, Martigues
  - Private Practice of Dr. Alain Boye, Nantes
  - Private Practice of Dr. Francois Volny, Nantes
  - Private Practice of Dr. Thierry Schaupp, Vihiers
- Germany (10):
  - Private Practice of Dr. Josef Junggeburth, Bad Wörishofen
  - Charite Campus Mitte, Universitatsmedizin Berlin, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - Private Practice of Dr. Isabelle Schenkenberger, Berlin
  - Private Practice of Dr. Tobias Marsen, Cologne
  - PD Dr. med. Bernhard Winkelmann, Frankfurt
  - Clinical Research Hamburg, Hamburg
  - Dr. Med. Susanne Mindt-Prufert, Hamburg
  - Private Practice for Internal Medicine & Cardiology, Heidelberg
  - IFG-Institut fur Gesundheitsforderung GmbH, Rüdersdorf
- New Zealand (5):
  - Centre for Clinical Research and Effective Practice (CCRep), Auckland
  - Christchurch Hospital, Christchurch
  - Greenlane Clinical Centre, Greenlane
  - Cardiology Clinical Trial Unit, Hamilton
  - Tauranga Hospital, Tauranga
- Spain (2):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital General Universitario de Elche, Elche

REFERENCES:
- [Derived] Bakris GL, Lindholm LH, Black HR, Krum H, Linas S, Linseman JV, Arterburn S, Sager P, Weber M. Divergent results using clinic and ambulatory blood pressures: report of a darusentan-resistant hypertension trial. Hypertension. 2010 Nov;56(5):824-30. doi: 10.1161/HYPERTENSIONAHA.110.156976. Epub 2010 Oct 4. PMID 20921430
- See also: Related Info — http://www.gilead.com